CLINICAL TRIAL: NCT05835089
Title: Evaluation of Some-puberty Related Hormones Among Children and Adolescents With Chronic Kidney Diseases
Brief Title: Evaluation of Some Puberty-related Hormones Among Children and Adolescents With Chronic Kidney Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Heba Mohamed Ahmed, resident doctor at pediatrics department, Sohag University
Other Study IDs: Soh-Med-23-04-18MS
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Evaluation of Some Puberty-related Hormones Among Children and Adolescents With Chronic Kidney Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children and adolescents with chronic kidney diseases: The serum level of LH, FSH, prolactin, Testosterone (in boys), estradiol (in girls) and Kisspeptin levels will be measured for all the study participants.
  Interventions: Diagnostic Test: serum kisspeptin levels
- control group of patients: The serum level of LH, FSH, prolactin, Testosterone (in boys), estradiol (in girls) and Kisspeptin levels will be measured for all the study participants.
  Interventions: Diagnostic Test: serum kisspeptin levels

INTERVENTIONS:
Diagnostic Test: serum kisspeptin levels — Evaluation of the serum level of LH, FSH, prolactin, Testosterone (in boys), estradiol (in girls) and Kisspeptin levels
  Other Names: The serum level of LH, FSH, prolactin, Testosterone (in boys), estradiol (in girls)

SUMMARY:
Puberty is the process of transition from childhood into adolescence, signaling the readiness of the human body for reproduction. The Hypothalamic-Pituitary Gonadotropin axis plays the primary role in initiating the puberty, where the hypothalamus secrets gonadotropin releasing hormone (GnRH) in a pulsatile manner, which in turn stimulates the release of luteinizing hormone (LH), and follicle stimulating hormone (FSH) from the anterior lobe of the pituitary gland, and in a final step these hormones stimulate the gonads to release their sex hormones (Testosterone and Estradiol) .

Chronic illnesses can affect this physiological process resulting in delayed puberty . Delayed puberty is defined as the lack of pubertal signs until the age of 13 years in girls, and the age of 14 years in boys. Delayed puberty is classified into two categories according to their cause; central gonadotropin deficiency (hypogonadotropic hypogonadism) and this type comprises delayed puberty due to chronic illness, while the second category of delayed puberty is due to gonadal disorders (hypergonadotropic hypogonadism).

Delayed puberty is common among pediatric patients with chronic kidney disease (CKD) - where glomerular filtration rate (GFR) is less than 60 ml/min per 1.73 m2. Previous studies suggested that, the cyclic pattern of GnRH release is lost in patients with CKD resulting in impairment of gonadotropins secretion from the anterior pituitary gland. Multiple hormonal factors had been proposed to be responsible for the pubertal delay in patients with CKD, the most prominent of which is the increasing levels of prolactin, LH and GnRH (4). Prolactin normally inhibits the release of GnRH from hypothalamus thus inhibiting the initiation of puberty and it was found to increase in patients with CKD secondary to increased production, slightly decreased clearance and decreased responsiveness to the hypothalamic inhibition of prolactin secretion.

Furthermore, recent studies reported that the Kisspeptin protein play an important role in the regulation and control of normal puberty, As it was found that the Kisspeptin neurons (the rostral periventricular region of the third ventricle (RP3V) and arcuate nucleus (ARC), are found in close association with the GnRH releasing neurons in the hypothalamus suggesting that these neurons might play a crucial role in activating and restoring the pulsatile release of GnRH, It was also found that inactivating mutations of the gene encoding for kisspeptin were associated with hypogonadotropic hypogonadism.

ELIGIBILITY:
Inclusion Criteria:Children and Adolescents aged 8 to 18 years, diagnosed with CKD and attending the pediatric nephrology clinic and the pediatric dialysis unit at Sohag University Hospital will be included.

In addition, Age- and sex-matched controls will be included from children and adolescents attending the general pediatric clinic at Sohag University Hospital for acute non-serious illnesses.

-

Exclusion Criteria: Pediatric post-renal transplant recipients and patients receiving hormonal replacement therapy for endocrinopathies and cases with any other associated chronic illness will be excluded from the study.

-

Ages: 8 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children and Adolescents aged 8 to 18 years, diagnosed with CKD
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
The serum level of Kisspeptin levels | one year
  The serum level of Kisspeptin levels will be measured for all the study participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brook CG. Mechanism of puberty. Horm Res. 1999;51 Suppl 3:52-4. doi: 10.1159/000053162. PMID 10592444
- [Background] Pozo J, Argente J. Delayed puberty in chronic illness. Best Pract Res Clin Endocrinol Metab. 2002 Mar;16(1):73-90. doi: 10.1053/beem.2002.0182. PMID 11987900
- [Background] Levey AS, Eckardt KU, Tsukamoto Y, Levin A, Coresh J, Rossert J, De Zeeuw D, Hostetter TH, Lameire N, Eknoyan G. Definition and classification of chronic kidney disease: a position statement from Kidney Disease: Improving Global Outcomes (KDIGO). Kidney Int. 2005 Jun;67(6):2089-100. doi: 10.1111/j.1523-1755.2005.00365.x. PMID 15882252
- [Background] Holley JL. The hypothalamic-pituitary axis in men and women with chronic kidney disease. Adv Chronic Kidney Dis. 2004 Oct;11(4):337-41. PMID 15492969
- [Background] Harter CJL, Kavanagh GS, Smith JT. The role of kisspeptin neurons in reproduction and metabolism. J Endocrinol. 2018 Sep;238(3):R173-R183. doi: 10.1530/JOE-18-0108. PMID 30042117